CLINICAL TRIAL: NCT03456336
Title: Management of the Patent Ductus Arteriosus in Premature Infants Trial (PDA Trial)
Brief Title: Management of the PDA Trial
Acronym: PDA
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: NICHD Neonatal Research Network (Network)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NICHD-NRN-0059; UG1HD112079 (NIH); UG1HD112097 (NIH); UG1HD112100 (NIH)
Record Dates: First submitted 2018-02-19; First posted 2018-03-07 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2025-01

CONDITIONS: Infant, Premature; Patent Ductus Arteriosus; Infant, Newborn, Diseases; Patent Ductus Arteriosus After Premature Birth
MeSH Terms: conditions — Premature Birth; Ductus Arteriosus, Patent; Infant, Newborn, Diseases | interventions — Watchful Waiting

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Active Treatment Group (Active Comparator): Infants assigned to the active treatment group will receive indomethacin or ibuprofen per their local site usual care dosing and schedule if the infant has a sPDA. The choice of indomethacin or ibuprofen will be left to the center, however, infants may only receive one or the other.
  Interventions: Other: Active Treatment
- Expectant Management Group (Active Comparator): Infants assigned to the expectant management group will receive indomethacin or ibuprofen if cardiopulmonary compromise occurs.
  Interventions: Other: Expectant Management

INTERVENTIONS:
Other: Active Treatment — Infants assigned to the active treatment group will receive indomethacin or ibuprofen per their local site usual care dosing and schedule if the infant has a sPDA. The choice of indomethacin or ibuprofen will be left to the center, however, infants may only receive one or the other. If the infant receives both, it will be considered a protocol violation.
  Arms: Active Treatment Group
Other: Expectant Management — Infants assigned to the expectant management group will receive indomethacin or ibuprofen if cardiopulmonary compromise occurs.
  Arms: Expectant Management Group

SUMMARY:
Estimate the risks and benefits of active treatment versus expectant management of a symptomatic patent ductus arteriosus (sPDA) in premature infants.

DETAILED DESCRIPTION:
This is a pragmatic randomized multicenter, effectiveness study comparing active treatment of a symptomatic patent ductus arteriosus (sPDA) to expectant management. We hypothesize in premature infants with a sPDA, expectant management reduces the incidence proportion of death or BPD by 10% (from 50% to 40%) when compared to active treatment.

Participants with a sPDA allocated to the active treatment arm will receive intravenous administration of indomethacin or ibuprofen (depending on center preference). The decision to ligate will be left to the clinical team. Participants with a sPDA allocated to the expectant management arm will receive supportive care at the clinical team's discretion and will receive indomethacin/ibuprofen or ligation if the infant develops cardiopulmonary compromise. The decision to ligate will be left to the clinical team.

The primary endpoint for the study will be death or BPD (as assessed by the physiologic definition) at 36 weeks postmenstrual age (PMA).

ELIGIBILITY:
Inclusion Criteria:

* Postnatal age 48 hours -21 days
* Infant 22 0/7 to 28 6/7 weeks gestation at birth
* sPDA, as defined as:

  1. Mild, Moderate, or Severe Clinical Criteria with Small or Moderate size PDA on echocardiogram
  2. Mild or Moderate Clinical Criteria with Large PDA on echocardiogram

Exclusion Criteria:

* Cardiopulmonary compromise
* Known congenital heart disease (besides atrial septal defect or ventricular septal defect)
* Known pulmonary malformation (e.g. congenital lobar emphysema, congenital pulmonary adenomatous malformation)
* Any condition which, in the opinion of the investigator, would preclude enrollment

Ages: 48 Hours to 21 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 836 (Estimated)
Dates: Start 2019-02-22 (Actual); Primary Completion 2025-03-02 (Actual); Study Completion 2027-05-30 (Estimated)

PRIMARY OUTCOMES:
Death or Bronchopulmonary Dysplasia (BPD) at 36 weeks PMA | birth to 36 week postmenstrual age
  Death or BPD. BPD will be defined by the physiologic definition.

SECONDARY OUTCOMES:
Mortality at 36 weeks PMA | birth to 36 week postmenstrual age
  mortality assessed at 36 week postmenstrual age
Mortality before discharge | birth to 120 days of life
  mortality assessed prior to hospital discharge
Bronchopulmonary dysplasia - Physiological Test | birth to 36 week postmenstrual age
  BPD defined by the physiologic test of oxygen therapy
Bronchopulmonary dysplasia - NIH Consensus Definition | birth to 36 week postmenstrual age
  BPD defined by the NIH consensus definition of moderate or severe
Necrotizing Enterocolitis (NEC) at 36 weeks PMA | birth to 36 weeks post menstrual age
  Proven NEC, no surgery, Stages IIA, IIB, or IIIA AND proven, surgery, Stage IIIB
Retinopathy of Prematurity at 36 weeks PMA | birth to 36 weeks post menstrual age
  Stage 3 or worse in either eye AND as any intervention therapy-retinal ablation, scleral buckle/vitrectomy, avastin or other anti-VEGF drug
Receipt of therapies designed to close the PDA | birth to 120 days
  Defined as ligation or cardiac catheterization
Weight at 36 weeks PMA | birth to 36 weeks post menstrual age
  Weight assessed at 36 weeks post menstrual age
Height at 36 weeks PMA | birth to 36 weeks post menstrual age
  Height assessed at 36 weeks post menstrual age
Head Circumference at 36 weeks PMA | birth to 36 weeks post menstrual age
  Head Circumference assessed at 36 weeks post menstrual age

OTHER OUTCOMES:
Necrotizing Enterocolitis (NEC) at status (2 years) | 26 months corrected age
  Proven NEC, no surgery, Stages IIA, IIB, or IIIA AND proven, surgery, Stage IIIB
Retinopathy of Prematurity at status (2 years) | 26 months corrected age
  Stage 3 or worse in either eye AND as any intervention therapy-retinal ablation, scleral buckle/vitrectomy, avastin or other anti-VEGF drug
Weight at status (2 years) | 26 months corrected age
  Weight assessed at status (2 years)
Height at status (2 years) | 26 months corrected age
  Height assessed at status (2 years)
Head Circumference at status (2 years) | 26 months corrected age
  Head Circumference assessed at status (2 years)
Neurodevelopmental impairment (NDI) at status (2 years) | 26 months corrected age
  Severe NDI will be defined by any of the following: a BSID III cognitive score < 70, Gross Motor Functional (GMF) Level of 3-5, blindness (<20/200 vision) or profound hearing loss (inability to understand commands despite amplification); moderate NDI will be defined as a BSID III cognitive score 70-84 and either a GMF level of 2 or a hearing deficit requiring amplification to understand commands or unilateral blindness; mild NDI will be defined by a cognitive score 70-84, or a cognitive score ≥ 85 and any of the following: presence of a GMF level 1 or hearing loss not requiring amplification. Normal (no NDI) will be defined by a cognitive score ≥ 85 and absence of any neurosensory deficits.

CONTACTS AND LOCATIONS:
Locations (19):
- United States (19):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Stanford University, Palo Alto, California
  - Sharp Mary Birch Hospital for Women & Newborns, San Diego, California
  - Emory University, Atlanta, Georgia
  - Northwestern Lurie Children's Hospital of Chicago, Chicago, Illinois
  - University of Iowa, Iowa City, Iowa
  - University of Mississippi Medical Center - Children's of Mississippi, Jackson, Mississippi
  - University of New Mexico, Albuquerque, New Mexico
  - University of Rochester, Rochester, New York
  - RTI International, Durham, North Carolina
  - Duke University, Durham, North Carolina
  - Cincinnati Children's Medical Center, Cincinnati, Ohio
  - Case Western Reserve University, Rainbow Babies and Children's Hospital, Cleveland, Ohio
  - Research Institute at Nationwide Children's Hospital, Columbus, Ohio
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Brown University - Women and Infants Hospital of Rhode Island, Providence, Rhode Island
  - University of Texas Southwestern Medical Center at Dallas, Dallas, Texas
  - University of Texas Health Science Center at Houston, Houston, Texas
  - University of Utah, Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: Yes
Per NIH Data Sharing Plan
Supporting Information: Study Protocol, SAP

REFERENCES:
- [Derived] Laughon MM, Thomas SM, Watterberg KL, Kennedy KA, Keszler M, Ambalavanan N, Davis AS, Slaughter JL, Guillet R, Colaizy TT, Cotten CM, Dhawan MA, Bose CL, Talbert J, Smucny S, Benitz WE, Rysavy MA, Ohls RK, Baserga MC, DeMauro SB, Jaleel M, Jackson WM, Carlo WA, Puopolo KM, Hibbs AM, Katheria A, Sanchez PJ, D'Angio CT, Patel RM, Johnson BA, Chock VY, Bhatt AJ, Merhar SL, Moore R, Laptook AR, Ghavam S, Fuller J, Vyas-Read S, Kicklighter SD, Steinbrekera B, Anderson K, Reynolds AM, Wyckoff MH, Montoya C, Das A, Do B, Chang S, Higgins RD, Walsh MC; Eunice Kennedy Shriver National Institute of Child Health and Human Development Neonatal Research Network. Expectant Management vs Medication for Patent Ductus Arteriosus in Preterm Infants: The PDA Randomized Clinical Trial. JAMA. 2025 Dec 9:e2523330. doi: 10.1001/jama.2025.23330. Online ahead of print. PMID 41364689
- See also: NRN Website — http://neonatal.rti.org